CLINICAL TRIAL: NCT01799850
Title: The Impact of Actos Treatment of Diabetes on Glucose Transporters in Muscle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Tennessee State University (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Charles A. Stuart, Professor, Internal Medicine, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPNA 02-037A
Record Dates: First submitted 2012-03-20; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Type 2
Keywords: muscle; glucose transporters; GLUT4; GLUT5; Actos
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actos (Active Comparator): Actos 30 mg daily
  Interventions: Drug: Pioglitazone
- placebo (Placebo Comparator): double blind placebo controlled
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone 30 mg daily, pill, eight weeks, placebo randomly assigned
  Other Names: Actos or placebo
  Arms: Actos
Drug: placebo — placebo assigned randomly, double blind
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
Subjects with type 2 diabetes will be treated with Actos or placebo for eight weeks and needle biopsies of muscle will quantify changes in any of seven different glucose transport proteins in muscle.

DETAILED DESCRIPTION:
Twelve subjects with type 2 diabetes, with fair control on oral medication, will be recruited to participate in a randomized, double-blind, placebo-controlled study of the impact on muscle glucose transporter expression of the addition of the insulin-sensitizing agent, pioglitizone (Takeda Pharmaceuticals). Therapy with the active drug will be at 30 mg daily. The other oral medications will be adjusted downward if hypoglycemia occurs. Glycemic control will be monitored by at least twice daily home blood glucose monitoring, weekly telephone contacts, and follow-up visits to the ETSU/VAMC Clinical Research Unit (CRU) every two weeks. During the eight weeks of therapy, subjects will be instructed to maintain their weight and keep their dietary and exercise regimens unchanged. Muscle biopsies will be obtained before and at the end of eight weeks of therapy. Specimens will be assayed for GLUT1, GLUT3, GLUT4, GLUT5, GLUT8, GLUT11, and GLUT12 mRNA and protein content and the subcellular distribution of these proteins as described below. Peroxisome proliferator-activated receptor gamma (PPARgamma), a member of the ligand-activated nuclear hormone receptor superfamily (14), will be quantified in these specimens by immunoblot as described below.

This study design involving a randomized, double-blinded, placebo-controlled treatment regimen is needed to control for confounding variables causing changes in glucose transporter expression that may be erroneously attributed to the drug. These potential variables include close contact with the diabetes management team resulting in improved compliance with diet, exercise, medication, and monitoring and thus better glycemic control, weight loss, or improved fitness.

ELIGIBILITY:
Inclusion Criteria:

* diabetes, type 2
* HbA1c less than 8.5

Exclusion Criteria:

* insulin therapy
* renal insufficiency
* clinically apparent coronary disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2002-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
change in muscle glucose transporter expression | post eight weeks treatment
  immunoblots pre and post, placebo and Actos

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Stuart, MD, Principal Investigator — ETSU Quillen College of Medicine
Locations (1):
- ETSU Quillen College of Medicine, Johnson City, Tennessee, United States

REFERENCES:
- [Result] Stuart CA, Howell ME, Yin D. Overexpression of GLUT5 in diabetic muscle is reversed by pioglitazone. Diabetes Care. 2007 Apr;30(4):925-31. doi: 10.2337/dc06-1788. Epub 2007 Jan 24. PMID 17251278